CLINICAL TRIAL: NCT05492461
Title: Physician-assisted Dying in Mentally Ill Patients - Which Criteria Are Decisive? An Exploratory Study in the General Population and in the Medical Profession About Physician-assisted Dying in Somatic Versus Mental Illness in Switzerland
Brief Title: Physician-assisted Dying in Mentally Ill Patients - Which Criteria Are Decisive?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Psychiatric Hospital of the University of Basel (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Christian G. Huber, Chief Physician, Psychiatric Hospital of the University of Basel
Other Study IDs: KZS Seed Grant 11/20
Record Dates: First submitted 2022-07-05; First posted 2022-08-08 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Physician-Assisted Suicide
MeSH Terms: conditions — Suicide, Assisted

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Swiss Physicians: A group of approximately 10'000 physicians practicing in the cantons of Basel-Stadt, Basel-Landschaft, Aargau, Lucerne, Graubünden, Ticino and Vaud.
- General population of Switzerland: A group of 10,000 people from the general population including the three language regions (German, Italian, and French)

SUMMARY:
Physician-assisted dying (PAD) is currently a highly controversial topic in medical ethics and public debates worldwide. It poses a moral conflict between the ethical principle of respect for patient autonomy and the ethical principle of beneficence in the sense of preserving life. Switzerland gives higher weight to the former principle: Article 115 of the Swiss Penal Code (StGB) permits PAD, provided it is not performed for "selfish reasons", and thus, occupies a special role in international comparison. However, the Swiss federal law does not regulate who exactly is entitled to access PAD, and there is no universal agreement in the concerned professional societies. Additional uncertainty arises when not the wish for PAD of a somatically ill person but that of a mentally ill person is to be assessed. It is therefore important for Switzerland - but also internationally - to regulate PAD for the mentally ill. On the one hand, mentally ill persons must not be discriminated in their desire for PAD compared to somatically ill persons while at the same time, their vulnerability must be taken into account. On the other hand, treating physicians must be protected in their ethical integrity and need security when they have to decide on PAD-requests. With the present study, we aim at contributing to the discussion of PAD in mentally ill patients and, with the help of an online/telephone survey, provide insights of the current situation in Switzerland within the general population and in the medical profession. This study addresses the following research questions: What is the attitude of the general population towards the current Swiss Academy of Medical Sciences (SAMS) ethical guidelines? What is the attitude of medical professionals? To what extent does the public discussion reflect the current situation in clinical practice? Does the stigmatization of the mentally ill have an influence on the assessment of their wish to die, and if so, where do prejudices need to be reduced? The study thus aims to expand the scientific literature on this highly relevant, currently controversial topic.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for participants from the general population are: (1) between 18 and 65 years old, and (2) sufficient knowledge of German, Italian, or French. Medical professionals are included if they are registered in one of the cantons Basel-Stadt, Basel-Landschaft, Aargau, Lucerne, Graubünden, Ticino or Vaud. Physicians from all specialties are to be surveyed to be able to draw a comparison between the different medical professionals.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For this study, a survey of two groups is planned: a group of 10,000 people from the general population including the three language regions (German, Italian, and French) as well as a group of 10'000 physicians practicing in the cantons of Basel-Stadt, Basel-Landschaft, Aargau, Lucerne, Graubünden, Ticino and Vaud. In total, the sample thus comprises 20'000 individuals.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Degree of consent to physician-assisted dying in somatic versus mental illness | during the procedure
  The primary endpoint will be the degree of consent to physician-assisted dying depending on the type of illness (somatic vs. mental) as assessed on a 5-point Likert scale (1 = I disagree; 5 = I agree).

SECONDARY OUTCOMES:
Degree of consent to physician-assisted dying as a function of other factors | during the procedure
  Degree of consent to physician-assisted dying on a 5-point Likert scale (1 = I disagree; 5 = I agree) scale as a function of
  1. the intolerable suffering
  2. decision-making capacity
  3. the availability of therapeutic options
  4. the terminal nature of the illness
Positioning of the respondents to the SAMS criteria of 2004, 2018 and 2021. | during the procedure
  Positioning of the respondents to the SAMS criteria of 2004, 2018 and 2021 as measured through spontaneously expressed opinions in an open answer format in the context of a qualitative evaluation.
Correlation between the positioning of the respondents on the SAMS criteria of 2004, 2018, and 2021 and the evaluation of the case vignettes | during the procedure
  Positioning of the respondents on the SAMS criteria as well as the positioning on the case vignettes will be measured on a 5-point Likert scale (1 = I disagree; 5 = I agree). Correlations will be calculated using the participants' ratings on these scales.
Correlation between the degree of stigmatization and the assessment of physician-assisted dying. | during the procedure
  The degree of stigmatization will be measured using the Bogardus scale (Bogardus, 1925) as well as the Staff Attitude to Coercion Scale (SACS). The Bogardus and SACS scores range from 1 to 4, with 1 representing low degree of consent and 4 a high degree of consent. The assessment of physician-assisted dying is measured on a 5-point Likert scale (1 = I disagree; 5 = I agree). Correlations will be calculated using the participants' scores on the three scales mentioned.
Comparison of the primary and secondary endpoints between the two groups. | during the procedure
  The primary endpoint will be the degree of consent to physician-assisted dying depending on the type of illness (somatic vs. mental) as assessed on a 5-point Likert scale (1 = I disagree; 5 = I agree). The secondary endpoint are measured as mentioned in secondary outcome 2-5, and 7.
  Using the participants' scores on the different scales as indicated, correlations between the different endpoints will calculated to compare the primary and secondary endpoints.
Positioning of the respondents to the SAMS criteria of 2004, 2018 and 2021. | during the procedure
  Positioning of the respondents to the SAMS criteria of 2004, 2018 and 2021 as measured by the agreement or disagreement when presented SAMS criteria of 2004, 2018 and 2021 on a 5-point Likert scale (1 = I disagree; 5 = I agree)

REFERENCES:
- [Derived] Kowalinski E, Ziltener T, Staub S, Moeller J, Trachsel M, Schneeberger AR, Franke I, Lang UE, Huber CG. Physician assisted-dying in mentally and somatically ill individuals in Switzerland: Protocol for survey-based study. Front Psychiatry. 2022 Oct 28;13:987791. doi: 10.3389/fpsyt.2022.987791. eCollection 2022. PMID 36386979